CLINICAL TRIAL: NCT05511142
Title: Effectiveness of Endotracheal Intubation and Mask Ventilation Procedural Skills Training on Preclinical Student Using Modified Peyton's Four-Step Approach During COVID-19 Pandemic
Brief Title: Intubation and Ventilation Skill Training Using Modified Peyton's Four-Step Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aldy Heriwardito, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IndonesiaUAnes396
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic Peyton's Four-Step Approach (Experimental): Students followed offline training session of endotracheal intubation and mask ventilation procedural skills
  Interventions: Other: Classic Peyton's Four-Step Approach
- Modified Peyton's Four-Step Approach (Experimental): Students followed online training session of endotracheal intubation and mask ventilation procedural skills
  Interventions: Other: Modified Peyton's Four-Step Approach

INTERVENTIONS:
Other: Classic Peyton's Four-Step Approach — Instructor demonstrated endotracheal intubation and mask ventilation procedural skills directly to the preclinical students, followed by direct hands-on practice using manequin, ended with giving feedback to the students
  Arms: Classic Peyton's Four-Step Approach
Other: Modified Peyton's Four-Step Approach — Video tutorial of endotracheal intubation and mask ventilation were given to the students without explanation, followed by video tutorial making using manequin (without instructor) by the students which will be uploaded to Youtube
  Arms: Modified Peyton's Four-Step Approach

SUMMARY:
Endotracheal intubation and mask ventilation procedural skills are basic skills which have to be learnt by medical student and have to be practiced directly. However, during COVID-19 pandemic, offline training was difficult to be conducted and new specific learning method has not established yet. The study aims to assess the effectiveness of modified Peyton's four-step approach, which can be implemented through online training, compared to the classic Peyton's four-step approach in learning endotracheal intubation and mask ventilation procedural skills.

ELIGIBILITY:
Inclusion Criteria:

* Preclinical students of Faculty of Medicine Universitas Indonesia agreed to participate and signed the consent
* Preclinical students of Faculty of Medicine Universitas Indonesia registered to attend every training session of endotracheal intubation and mask ventilation under Basic Clinical Skills module
* 100% attendance in every session

Exclusion Criteria:

* Students who have attended endotracheal intubation and mask ventilation training beforehand
* Students who have learnt endotracheal intubation and mask ventilation under Basic Clinical Skills module beforehand

Drop out Criteria:

* Preclinical students of Faculty of Medicine Universitas Indonesia who quit from Basic Clinical Skills module during research
* Students who have never attended the training session

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Global rating | by the end of Basic Clinical Skill module, approximately 1-3 months after training
  numeric score
Actual mark | by the end of Basic Clinical Skill module, approximately 1-3 months after training
  numeric score

SECONDARY OUTCOMES:
Satisfaction score | by the end of Basic Clinical Skill module, approximately 1-3 months after training
  using Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Aldy Heriwardito, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided